CLINICAL TRIAL: NCT01991015
Title: Gender Differences in Inpatient Goals of Care Discussions in Patients With Advanced Cancer
Brief Title: Goals of Care Discussions for Hospitalized Patients With Advanced Cancer
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Rashmi Sharma, Assistant Professor of Medicine, Northwestern University
Other Study IDs: NU_STU00077507; K12HD055884 (NIH)
Record Dates: First submitted 2013-11-18; First posted 2013-11-25 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2015-02

CONDITIONS: Metastatic Cancer
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of this study is to better understand gender differences in end-of-life communication between physicians and patients with advanced cancer in the hospital.

ELIGIBILITY:
Inclusion Criteria:

* English speaking, have metastatic cancer that has progressed despite treatment

Exclusion Criteria:

* Cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients must be hospitalized at Northwestern Memorial Hospital and be having a goals of care discussion with their physician. In addition, eligible patients must be greater than the age of 18 years, speak English fluently, be able to physically and cognitively complete the informed consent process, and have metastatic cancer that has progressed despite treatment.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2013-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Quality of end-of-life communication | 15 months
  This is a qualitative study and the outcome will be assessed by coding the transcripts of the goals of care discussions. We will use the Roter Interaction Analysis System (RIAS) in which coders assign 1 of 37 mutually exclusive and exhaustive categories to each complete thought expressed (referred to as an utterance). Utterances are combined to reflect "instrumental" (e.g., biomedical exchange, psychosocial exchange, and partnership building) and "affective" behaviors (e.g., social conversation, positive and negative statements, and emotional statements). Additional global measures include patient-centeredness, verbal dominance, and tone.

CONTACTS AND LOCATIONS:
Overall Officials: Rashmi K Sharma, MD, MHS, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States